CLINICAL TRIAL: NCT03570697
Title: High-Resolution Assessment of Coronary Plaques in a Global Evolocumab Randomized Study (HUYGENS)
Brief Title: Imaging of Coronary Plaques in Participants Treated With Evolocumab
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20160184; 2017-003236-37 (EudraCT Number)
Record Dates: First submitted 2018-06-18; First posted 2018-06-27 (Actual); Results first posted 2021-11-24 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Coronary Artery Disease (CAD)
Keywords: Optical coherence tomography (OCT); Intravascular ultrasound (IVUS); Coronary angiography; Coronary artery disease; Cardiovascular events; Coronary atherosclerotic plaques; Lipid-lowering therapy; Statin; Maximally tolerated statin therapy
MeSH Terms: conditions — Coronary Artery Disease | interventions — evolocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a double-blind study. Treatment assignment will be blinded to all subjects, site personnel, and Amgen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Evolocumab (Experimental): Participants receive evolocumab subcutaneous injection once every month (QM) for 48 weeks. As prescribed and provided by the investigator, participants will be treated with maximally tolerated statin therapy, not expected to change for the duration of the study participation.
  Interventions: Drug: Evolocumab; Drug: Statin therapy
- Placebo (Placebo Comparator): Participants receive placebo subcutaneous injection QM for 48 weeks. As prescribed and provided by the Investigator, participants will be treated with maximally tolerated statin therapy, not expected to change for the duration of the study participation.
  Interventions: Drug: Placebo; Drug: Statin therapy

INTERVENTIONS:
Drug: Evolocumab — Participants will receive evolocumab (AMG 145) subcutaneous monthly.
  Other Names: Repatha, AMG 145, EvoMab
  Arms: Evolocumab
Drug: Placebo — Participants will receive matching placebo subcutaneous monthly.
  Arms: Placebo
Drug: Statin therapy — high-intensity statin treatment with atorvastatin ≥ 40 mg daily or equivalent as background therapy
  Investigators will up-titrate statin therapy to the maximally tolerated dose, in accordance with local guidelines, prior to randomization.

SUMMARY:
To evaluate the effect of evolocumab on fibrous cap thickness (FCT) in participants with non-ST-elevation acute coronary syndrome (NSTE-ACS) who are taking maximally tolerated statin therapy.

DETAILED DESCRIPTION:
This study seeks to identify morphologic changes, such as increase in FCT in atherosclerotic plaques associated with treatment with evolocumab and maximally tolerated statin therapy with or without additional lipid-modifying medication in patients presenting with NSTE-ACS using optical coherence tomography (OCT; primary, secondary, and exploratory endpoints).

ELIGIBILITY:
Inclusion Criteria:

* Provided informed consent prior to initiation of any study-specific activities/procedures.
* Age greater than or equal to 18 years at screening
* Clinical indication for coronary angiography during admission due to NSTE-ACS with interventional treatment of culprit plaque
* An eligible low-density lipoprotein cholesterol (LDL-C) level via local lab assessment based on statin use at screening

No statin use: greater than or equal to 130 mg/dL Low- or moderate-intensity statin use greater than or equal to 80 mg/dL High-intensity statin use greater than or equal to 60 mg/dL

* On maximally tolerated statin therapy in accordance with standard of care per local guidelines prior to randomization.
* Tolerates placebo run-in injection at screening
* Meets all the following criteria at the qualifying coronary angiogram:

Angiographic evidence of coronary artery disease (CAD) with greater than or equal to 20% reduction of lumen diameter by angiographic visual estimation, in addition to the culprit plaque.

Left main coronary artery must not have a greater than 50% reduction in lumen diameter by visual angiographic estimation.

Targeted vessel:

May not be the culprit vessel for the current or a previous myocardial infarction (MI).

Has not undergone prior percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG), and may not be a bypass graft.

May not be a candidate for PCI or CABG currently or over the next 12 months, in the opinion of the investigator.

Must be accessible by the optical coherence tomography (OCT) catheter.

Targeted segment:

Must have up to 50% but not greater than 50% reduction in lumen diameter by visual angiographic estimation and must be at least 40 mm in length.

Must contain at least 1 image with a fibrous cap thickness (FCT) of less than or equal to 120 μm and at least 1 image with a lipid arc of greater than 90° as determined by the imaging core laboratory Distal plaques of up to 50% stenosis by visual angiographic estimation are permitted, provided that such stenosis is not a target for PCI or CABG.

Exclusion Criteria:

* ST-segment elevation myocardial infarction (STEMI) or left bundle branch block (LBBB).
* Acute coronary syndromes (ACS) likely to be caused by a non-atherosclerotic process, in the opinion of the investigator (ie, type 2 myocardial infarction, which is characterized by an imbalance between myocardial oxygen demand and supply).
* Clinically significant heart disease which in the opinion of the investigator is likely to require coronary bypass surgery, PCI (does not apply to PCI of non-STEMI (NSTEMI) during initial screening angiogram), surgical or percutaneous valve repair and/or replacement during the course of the study.
* Any cardiac surgery within 6 weeks prior to screening.
* Triglycerides greater than or equal to 400 mg/dL (4.5 mmol/L) at screening.
* Moderate to severe renal dysfunction, defined as an estimated glomerular filtration rate (eGFR) less than 30 mL/min/1.73m^2 at screening.
* Malignancy except non-melanoma skin cancers, cervical, or breast ductal carcinoma in situ within the last 5 years.
* Intolerant to statins as determined by principal investigator.
* Previously received or receiving evolocumab or any other therapy to inhibit proprotein convertase subtilisin/kexin type 9 (PCSK9).
* Previously received a cholesterol ester transfer protein (CETP) inhibitor (ie, anacetrapib, dalcetrapib, evacetrapib), mipomersen, lomitapide, or has undergone LDL-apheresis in the last 12 months prior to LDL-C screening.
* Currently receiving treatment in another investigational device or drug study, or less than 30 days since ending treatment on another investigational device or drug study(ies). Other investigational procedures while participating in this study are excluded.
* Baseline OCT does not meet OCT imaging criteria as determined by the imagine core laboratory technical standards.
* Female subject is pregnant or breastfeeding or planning to become pregnant or breastfeed during treatment and for an additional 15 weeks after the last dose of investigational product. (Females of childbearing potential should only be included in the study after a confirmed menstrual period and a negative highly sensitive urine or serum pregnancy test.)
* Female subjects of childbearing potential unwilling to use 1 acceptable method of effective contraception during treatment and for an additional 15 weeks after the last dose of investigational product.
* Female subject who has not used an acceptable method(s) of birth control for at least 1 month prior to screening, unless the female subject is sterilized or postmenopausal.
* Known sensitivity to any of the products or components (eg, carboxymethylcellulose) to be administered during dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2021-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (33):
- United States (5):
  - University of California at Los Angeles, Los Angeles, California
  - Medstar Heart and Vascular Institute, Washington D.C., District of Columbia
  - Midwest Cardiovascular Research And Education Foundation, Elkhart, Indiana
  - Saint Louis University Hospital, St Louis, Missouri
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
- Australia (5):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - The Northern Hospital, Epping, Victoria
- Czechia (2):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
- Germany (3):
  - Charite UniversitÃ¤tsmedizin Berlin Campus Benjamin Franklin, Berlin
  - UniversitÃ¤res Herzzentrum Hamburg GmbH, Hamburg
  - Deutsches Herzzentrum MÃ¼nchen des Freistaates Bayern, MÃ¼nchen
- Hungary (4):
  - Allami Szivkorhaz Balatonfured, Balatonfüred
  - Semmelweis Egyetem, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
- Italy (7):
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII, Bergamo
  - Azienda Ospedaliera Santa Croce e Carle, Cuneo
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - IRCCS Centro Cardiologico Monzino, Milan
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Azienda Ospedaliera San Giovanni Addolorata, Roma
  - IRCCS Istituto Clinico Humanitas, Rozzano MI
- Netherlands (7):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Vrjie Universiteit Medisch Centrum, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Radboud Universitair Medisch Centrum, Nijmegen
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen
  - Elisabeth-TweeSteden Ziekenhuis, Tilburg
  - Isala Klinieken, Zwolle

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Nicholls SJ, Nissen SE, Prati F, Windecker S, Kataoka Y, Puri R, Hucko T, Kassahun H, Liao J, Somaratne R, Butters J, Di Giovanni G, Jones S, Psaltis PJ. Assessing the impact of PCSK9 inhibition on coronary plaque phenotype with optical coherence tomography: rationale and design of the randomized, placebo-controlled HUYGENS study. Cardiovasc Diagn Ther. 2021 Feb;11(1):120-129. doi: 10.21037/cdt-20-684. PMID 33708484
- [Background] Pharmacoeconomic Review Report: Icosapent Ethyl (Vascepa): (HLS Therapeutics Inc.): Indication: Prevention of cardiovascular events in statin-treated patients [Internet]. Ottawa (ON): Canadian Agency for Drugs and Technologies in Health; 2020 Aug. Available from http://www.ncbi.nlm.nih.gov/books/NBK566010/ PMID 33355725
- [Derived] Di Giovanni G, Fujino M, Kataoka Y, Butters J, Hucko T, Puri R, Nissen SE, Nelson AJ, Psaltis PJ, Nicholls SJ. Impact of evolocumab on plaque phenotypic changes in patients with acute coronary syndrome and elevated lipoprotein(a) levels: a HUYGENS secondary analysis. Eur J Prev Cardiol. 2025 Apr 8:zwaf211. doi: 10.1093/eurjpc/zwaf211. Online ahead of print. PMID 40424182
- [Derived] Fujino M, Di Giovanni G, Butters Bhsc J, Kataoka Y, Hucko T, Nelson AJ, Nissen SE, Psaltis PJ, Nicholls SJ. Achieved levels of apolipoprotein B and plaque composition after acute coronary syndromes: Insights from HUYGENS. Atherosclerosis. 2025 Apr;403:119145. doi: 10.1016/j.atherosclerosis.2025.119145. Epub 2025 Feb 20. PMID 40020597
- [Derived] Nicholls SJ, Kataoka Y, Nissen SE, Prati F, Windecker S, Puri R, Hucko T, Aradi D, Herrman JR, Hermanides RS, Wang B, Wang H, Butters J, Di Giovanni G, Jones S, Pompili G, Psaltis PJ. Effect of Evolocumab on Coronary Plaque Phenotype and Burden in Statin-Treated Patients Following Myocardial Infarction. JACC Cardiovasc Imaging. 2022 Jul;15(7):1308-1321. doi: 10.1016/j.jcmg.2022.03.002. Epub 2022 Mar 16. PMID 35431172
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 23 research centers in Australia (2), Czech Republic (2), Germany (2), Hungary (4), Italy (6), and the Netherlands (7), from November 2018 to December 2019.
Pre-assignment Details: Participants were randomized 1:1 into 2 treatment groups: evolocumab 420 mg subcutaneously (SC) monthly (QM) or placebo SC QM.
  Randomization was stratified by current statin use (> 4 weeks or ≤ 4 weeks) at screening.
Groups:
- Placebo: Placebo SC injection QM for 48 weeks. Background maximally tolerated statin therapy for the duration of the study participation.
- Evolocumab: Evolocumab 420 mg SC injection QM for 48 weeks. Background maximally tolerated statin therapy for the duration of the study participation.
Period: Overall Study
Arm/Group | Placebo | Evolocumab
Started | 82 | 82
Received at Least 1 Dose of Study Drug | 81 | 80
Completed | 76 | 79
Not Completed | 6 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 2 | 0
Not completed — Withdrawal by Subject | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Evolocumab | Total
Number analyzed (Participants) | 82 | 82 | 164
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (9.4) | 61.1 (10.0) | 60.8 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 20 | 46
  Male | 56 | 62 | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 81 | 78 | 159
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 2
  White | 80 | 79 | 159
  Other, Not Specified | 1 | 2 | 3
Stratification Factor: Statin Use at Screening [Count of Participants; unit: Participants]
  > 4 weeks of statin use | 20 | 19 | 39
  ≤ 4 weeks of statin use | 62 | 63 | 125
Minimum Fibrous Cap Thickness (FCT) [Mean (Standard Deviation); unit: µm] — Minimum FCT as determined by optical coherence tomography (OCT). Minimum FCT for a participant is defined as the minimum of all minimum FCT measurements within each individual frame across all frames of that participant. Higher value of FCT indicates a better situation. Population: Full Analysis Set: all participants who received at least 1 dose of study drug.
  µm
    number analyzed (Participants) | 81 | 80 | 161
    (all) | 54.6 (15.1) | 56.6 (17.8) | 55.6 (16.5)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Minimum FCT
Description: Absolute change from baseline in minimum FCT in a matched segment of artery as determined by OCT. Minimum FCT for a participant is defined as the minimum of all minimum FCT measurements within each individual frame across all frames of that participant. Higher value of FCT indicates a better situation.
Time Frame: Baseline, week 50
Population: Full Analysis Set: all participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: µm
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 81 | 80
µm | 21.5 (5.2) | 42.7 (5.1)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority; p = 0.015, ANCOVA; Treatment difference = 21.2, 95% CI 2-sided [4.7 to 37.7], Standard Error of Mean 7.9

2. Secondary Outcome: Percent Change From Baseline in Minimum FCT
Description: Percent change from baseline in minimum FCT in a matched segment of artery as determined by OCT. Minimum FCT for a participant is defined as the minimum of all minimum FCT measurements within each individual frame across all frames of that participant. Higher value of FCT indicates a better situation.
Time Frame: Baseline, week 50
Population: Full Analysis Set: all participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 81 | 80
percent change | 44.30 (11.76) | 81.76 (10.94)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority; p = 0.041, ANCOVA; Treatment difference = 37.47, 95% CI 2-sided [1.63 to 73.31], Standard Error of Mean 17.04

3. Secondary Outcome: Absolute Change From Baseline in Mean Minimum FCT
Description: Absolute change from baseline in mean minimum FCT for all images assessed in an individual participant as determined by OCT. Minimum FCT for a participant is defined as the minimum of all minimum FCT measurements within each individual frame across all frames of that participant. Higher value of FCT indicates a better situation.
Time Frame: Baseline, week 50
Population: Full Analysis Set: all participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: µm
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 81 | 80
µm | 29.78 (6.88) | 62.29 (5.95)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority; p = 0.003, ANCOVA; Treatment difference = 32.51, 95% CI 2-sided [12.67 to 52.35], Standard Error of Mean 9.52

4. Secondary Outcome: Absolute Change From Baseline in the Maximum Lipid Arc
Description: Absolute change from baseline in the maximum lipid arc in a matched segment of artery as determined by OCT. Lower value of lipid arc indicates a better situation.
Time Frame: Baseline, week 50
Population: Full Analysis Set: all participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: degrees
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 81 | 80
degrees | -31.4 (9.0) | -57.5 (7.4)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority; p = 0.032, ANCOVA; Treatment difference = -26.0, 95% CI 2-sided [-49.6 to -2.4], Standard Error of Mean 11.4

5. Secondary Outcome: Absolute Change From Baseline in Minimum FCT in Lipid Rich Plaques
Description: Absolute change from baseline in minimum FCT in lipid rich plaques as determined by OCT. Lipid rich plaques are defined as minimum FCT less than 120 μm and lipid arc greater than 90° in at least 3 consecutive images as determined by OCT. Higher value of FCT indicates a better situation
Time Frame: Baseline, week 50
Population: Full Analysis Set: all participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: μm
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 81 | 80
μm | 24.6 (5.5) | 40.6 (5.5)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority; p = 0.036, ANCOVA; Treatment difference = 16.0, 95% CI 2-sided [1.1 to 31.0], Standard Error of Mean 7.5

6. Secondary Outcome: Absolute Change From Baseline in Maximum Lipid Arc in Lipid Rich Plaques
Description: Absolute change from baseline in maximum lipid arc in lipid rich plaques. Lipid rich plaques are defined as minimum FCT less than 120 μm and lipid arc greater than 90° in at least 3 consecutive images as determined by OCT. Lower value of lipid arc indicates a better situation.
Time Frame: Baseline, week 50
Population: Full Analysis Set: all participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: degrees
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 81 | 80
degrees | -31.9 (8.1) | -61.9 (7.9)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority; p = 0.005, ANCOVA; Treatment difference = -30.0, 95% CI 2-sided [-50.5 to -9.5], Standard Error of Mean 10.4

7. Secondary Outcome: Absolute Change From Baseline in Lipid Core Length in Lipid Rich Plaques
Description: Absolute change from baseline in lipid core length in lipid rich plaques. Lipid rich plaques are defined as minimum FCT less than 120 μm and lipid arc greater than 90° in at least 3 consecutive images as determined by OCT. Lower value of lipid core length indicates a better situation.
Time Frame: Baseline, week 50
Population: Full Analysis Set: all participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 81 | 80
mm | -3.33 (0.64) | -5.76 (0.61)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority; p = 0.003, ANCOVA; Treatment difference = -2.43, 95% CI 2-sided [-4.04 to -0.82], Standard Error of Mean 0.81

ADVERSE EVENTS:
Time Frame: All cause mortality reporting period is from the 1st dose of investigational product (IP) up to the end of study (EOS) date (Week 52). Adverse event (AE) reporting period is from the 1st dose of IP up to and including 30 days after the last dose of IP date or the EOS date (Week 52) whichever is earlier.
Description: Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug. All-cause mortality is reported for all participants randomized.
Arm/Group | Placebo | Evolocumab
All-Cause Mortality (participants affected / at risk) | 2/82 | 0/82
Serious Adverse Events (participants affected / at risk) | 16/81 | 13/80
Other Adverse Events (participants affected / at risk) | 30/81 | 31/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=81) | Evolocumab (N=80)
Normocytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 3 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Enterococcal infection (Infections and infestations) | 0 | 1
Meningitis staphylococcal (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Carotid artery restenosis (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 1
Pulmonary hypertensive crisis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=81) | Evolocumab (N=80)
Angina pectoris (Cardiac disorders) | 7 | 4
Bradycardia (Cardiac disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 4 | 3
Fatigue (General disorders) | 2 | 3
Non-cardiac chest pain (General disorders) | 0 | 2
Influenza (Infections and infestations) | 2 | 1
Pneumonia (Infections and infestations) | 0 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2
Glucose tolerance impaired (Metabolism and nutrition disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 5
Headache (Nervous system disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Drug eruption (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Hypertension (Vascular disorders) | 5 | 6
Hypotension (Vascular disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2018-04-19): https://cdn.clinicaltrials.gov/large-docs/97/NCT03570697/Prot_002.pdf
  • Statistical Analysis Plan (2021-01-15): https://cdn.clinicaltrials.gov/large-docs/97/NCT03570697/SAP_001.pdf